CLINICAL TRIAL: NCT01052935
Title: A Phase I Extension Study to Assess the Long-Term Persistence of GBS Serotype Ia Antibodies in Women Previously Immunized With a GBS Ia Crm-Glycoconjugate Vaccine
Brief Title: A Study to Assess the Persistence of a GBS Antibody in Women Previously Immunized With a GBS Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V98P1E1
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Group B Streptococcus (GBS) Disease
Keywords: Group B streptococcus; GBS; Vaccine
MeSH Terms: conditions — Guillain-Barre Syndrome; Disease | interventions — Vaccines

ARMS (1):
- Arm 1 (No Intervention): This is a phlebotomy study.
  Interventions: Biological: Group B streptococcus (GBS) vaccine

INTERVENTIONS:
Biological: Group B streptococcus (GBS) vaccine — No vaccine will be administered in this study. Only one study visit is required.
  Subjects will return to the clinic for a single visit at 24 months (± 3 months) after the last injection administered in the V98P1 study.

SUMMARY:
This study looks at the body's immune responses to a GBS vaccine 2 years after the orginal vaccine(s) were given in the V98P1 study. Blood will be drawn and evaluated for GBS antibody levels.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have given written consent.
* Individuals who participated in V98P1 and received the complete schedule of vaccinations.

Exclusion Criteria:

* Individuals who have not given written consent.
* Subjects who did not receive the complete schedule of vaccination in V98P1.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2010-01 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Antibody (Ab) response data at 24-months after the last injection given in study V98P1 GMCs, GMRs and associated 95% confidence intervals will also be determined | 24- months post last injection from V98P1

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Pharmacokinetic and Analytical Studies, Via Mastri, 36, CH - 6853 Ligornetto, Switzerland